CLINICAL TRIAL: NCT04354090
Title: Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of JY09, a Long-acting Glucagon-like Peptide-1 Mimetic, in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of JY09
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Dongfang Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: DFBT-JY09-101a
Record Dates: First submitted 2020-04-14; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 0.3-mg (Experimental): Eligible subjects received 0.3 mg placebo or JY09 on day 1 in this cohort
  Interventions: Drug: JY09
- Cohort 0.7-mg (Experimental): Eligible subjects received 0.3 mg placebo or JY09 on days 1, and 0.7 mg placebo or JY09 on days 22
  Interventions: Drug: JY09
- Cohort 1.5-mg (Experimental): Eligible subjects received 0.7 mg placebo or JY09 on days 1, and 1.5 mg placebo or JY09 on days 22
  Interventions: Drug: JY09
- Cohort 3.0-mg (Experimental): Eligible subjects received 0.7 mg placebo or JY09 on days 1, and 3.0 mg placebo or JY09 on days 22
  Interventions: Drug: JY09
- Cohort 6.0-mg (Experimental): Eligible subjects received 0.7 mg placebo or JY09 on days 1, and 1.0 mg placebo or JY09 on days 15, and 6.0 mg placebo or JY09 on days 30
  Interventions: Drug: JY09

INTERVENTIONS:
Drug: JY09 — Subcutaneous injection
  Other Names: Placebo

SUMMARY:
JY09 is a glucagon-like peptide-1 (GLP-1) mimetic generated by genetic fusion of a Exendin-4 dimer to human immunoglobulin Fc.

In this Double-blind, randomized, placebo-controlled trial, 41 healthy subjects received placebo or escalating doses of JY09 on day 1 in the first cohort, and on days 1 and 22 in the following sequential cohort 2-4, and on days 1, 15, and 30 in the cohort 5: cohort 1: 0.3 mg; cohort 2: 0.3 + 0.7 mg; cohort 3: 0.7+1.5 mg; cohort 4: 0.7+3.0 mg; and cohort 5: 0.7 + 1.5 + 6.0 mg. The primary endpoints were the incidence of adverse events and serious adverse events related to JY09. Secondary endpoints included pharmacodynamics and pharmacokinetics parameters, as well as anti-JY09 antibody incidence and titers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Male's mass is ≥50 kg, female's mass is ≥45 kg, have a body mass index between 18 and 26 kg/m^2
* Subjects or their legal representative signed informed consent
* agree to use instruments of contraception from the time of the first dose until 6 months after the last dose of investigational drug, avoid pregnancy make yourself or your mate
* Able to keep good communication with investigator and comply with the requirements of the clinical trials

Exclusion Criteria:

* Smokers,quitting time less than 3 months , or can't quit smoking during the trial
* Use of any prescription drugs within 4 weeks prior dosing, or over-the-counter medication (vitamins, herbal supplements, dietary supplements) within 2 weeks prior to dosing,or being treated for a direct lower gastrointestinal or using steroids
* Participation in any clinical investigation within 3 months prior to dosing
* Donation or loss of 400 mL or more of blood within 8 weeks prior to first dosing
* Significant illness within 2 weeks prior to dosing,and investigator judge doesn't fit to participate in this trial
* A history of clinical significance of abnormal ECG
* A history of diabetes, hyperuricemia and hyperlipidemia
* A history of acute or chronic bronchial spasms
* Have clinical significant gastrointestinal diseases
* Have serious, progressive, or uncontrolled organ or system diseases
* Abuse of drug or alcohol within 12 months before first dosing
* People who are pregnant, nursing mothers, or in the near future plan to be pregnant,or show pregnancy test positive before into group
* Subjects who, in the opinion of the investigator, are in any way unsuitable to participate in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2019-06-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events related to JY09 | Up to day 21

SECONDARY OUTCOMES:
Pharmacodynamics parameters: Cmax | Up To day 42
  Average Cmax of each dose level
Pharmacodynamics parameters: AUC | Up to day 42
  Average AUC follewing single dose of each doase level
Pharmacodynamics parameters: Half-life | Up to day 42
  Average Half-life of each dose level
Pharmacokinetics parameters | Day 5
  OGTT test was conducter predose and 5 days after the target dose in each cohorts
Immunogenicity | Up To day 42
  Anti-JY09 antibody incidence at each dose level

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li, M.D., Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No